CLINICAL TRIAL: NCT01981226
Title: Sonoelastographic Changes After Low Energy Extracorporeal Shock Wave Therapy (ESWT) in Plantar Fasciitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Sonoelastographic Changes After Low Energy Extracorporeal Shock Wave Therapy (ESWT) in Plantar Fasciitis, National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201007055R
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar

ARMS (1):
- Extracoporeal shock wave (Experimental): Extracoporeal shock wave, 3000 shots/time, once a week for 3 weeks, treatment duration:30 minutes/time, shock wave freqency：2-4Hz, energy level:0.8-1.0 mJ/mm2
  Interventions: Device: Extracoporeal shock wave

INTERVENTIONS:
Device: Extracoporeal shock wave — Extracoporeal shock wave, 3000 shots/time, once a week for 3 weeks, treatment duration:30 minutes/time, shock wave freqency：2-4Hz, energy level:0.8-1.0 mJ/mm2

SUMMARY:
Extracoporeal shock wave therapy(ESWT) was perfomed on the plantar fascia of chornic plantar fasciitis patients. Pre-ESWT and post-ESWT pain intensity, sonography and sonoelastrography of the plantar fascia was checked. Our hypothesis is that the plantar fascia stiffness increased after ESWT as clinical symptom improves.

DETAILED DESCRIPTION:
For patient who met the inclusion criteria, we check sonography and sonoelastography for their plantar fascias and obtain a thorough evulation questionaire for clinical symptom and pain condition and intensity in various conditions, also SF-36 questionaire first. Inform consent was done.

After the ESWT, we follow patient with questionaire and sonography/sonoelastography at 1-week, 1-month, 3-month, 6-month, 9-month, and 12-month post-ESWT time.

The colored sonoelastographic image was analysed by computer software "Image-J" with hue analysis method and relative stiffness of selected area within proximal plantar fascia wasa obtained for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* pain for more than 6 months，poor response to the conservative treatments
* Sonography showed plantar fasciitia>4.0mm)

Exclusion Criteria:

* Acute infection of soft tissue/bone
* Malignant primary disease
* Blood coagulation disorders
* Pregnancy
* Patients with pacemaker
* foot deformity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-09; Primary Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Sonoelastographic changes of plantar fascia after ESWT | pre-treatment, 1 week, 1 month, 3 month, 6 month, 9 month, 12 month

SECONDARY OUTCOMES:
Plantar fascia thickness | pre-treatment, 1 week, 1 month, 3 month, 6 month, 9 month, 12 month

OTHER OUTCOMES:
Pain intensity(VAS scale) | pre-treatment, 1 week, 1 month, 3 month, 6 month, 9 month, 12 month

CONTACTS AND LOCATIONS:
Locations (1):
- Natinal Taiwan University Hospital, Taipei, Taiwan, Taiwan